CLINICAL TRIAL: NCT06581796
Title: Examination of the Maternal Serum Pepsinogen-1 in Patients Diagnosed With Severe Hyperemesis Gravidarum: A Prospective Case-control Study
Brief Title: Pepsinogen-1 Serum Levels in Hyperemesis Gravidarum
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Fahri Burcin Firatligil, Specialist doctor in obstetrics and gynecology and Fellow student in Perinatology, Ankara Etlik City Hospital
Other Study IDs: AECH-FIRATLIGIL-002
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Hyperemesis Gravidarum; Pregnant With Complication
Keywords: Pepsinogen; Hyperemesis; Pregnancy
MeSH Terms: conditions — Hyperemesis Gravidarum; Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — Singleton nulliparous pregnant women who had been diagnosed with hyperemesis gravidarum in first trimester had blood samples taken at 8:00 am on the first visit to the outpatient clinic after an 8-hour fasting state
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: pregnant women with hyperemesis gravidarum
  Interventions: Other: pepsinogen-1
- Control group: pregnant women without hyperemesis gravidarum
  Interventions: Other: pepsinogen-1

INTERVENTIONS:
Other: pepsinogen-1 — association between pepsinogen 1 serum level with hyperemesis gravidarum

SUMMARY:
In this study, the investigators planned to investigate maternal serum pepsinogen-1 (MSPG-1) levels in pregnant women with severe hyperemesis gravidarum (HG) and pregnant women without severe HG.

HG is the most common cause of hospitalization in the first trimester of pregnancy and represents an economic burden on the healthcare system. Therefore, our aim in this study was to investigate whether there is a statistical difference in MSPG-1 levels between pregnant women with severe HG and pregnant women without severe HG and to determine a cut-off value for MSPG-1 levels for the indication of hospitalization of pregnant women with HG.

The study poses no risk to the pregnant woman or the fetus.

DETAILED DESCRIPTION:
The study will enroll pregnant women in the first trimester with maternal age between 21 and 35 years who were diagnosed with hyperemesis gravidarum and had no fetal congenital or chromosomal abnormalities and who were admitted to the perinatology outpatient clinic of Etlik City Hospital. The investigators will include 40 cases with no signs and diagnosis of systemic maternal disease and no chronic drug use as a case group and 40 healthy pregnant women matched for age, gestational week and body mass index as a control group.

ELIGIBILITY:
Inclusion Criteria:

* A singleton pregnancy
* Between 21 and 35 years old
* Diagnosis of hyperemesis gravidarum

Exclusion Criteria:

* Multiple pregnancy
* Fetal congenital and chromosomal abnormalities
* Chronic drug use, alcohol and smoking
* Pregnant women with diabetes or obesity, peptic ulcer or gastritis, liver and/or gallbladder disease (cholangitis or gallstones), thyroid dysfunction, urinary tract infection, celiac disease, cardiovascular or renal disease

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: The singleton pregnant women who were diagnosed with hyperemesis gravidarum were included in the study group (group I) and the singleton pregnant women who had a healthy pregnancy were included in the control group (group II). For each pregnant woman who met the inclusion and exclusion criteria and was eligible for Group I, the first patient in the ranking order of the files who met the criteria previously mentioned in the Materials and Methods section was selected for Group II.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Pepsinogen-1 serum level | between 5 and 14 weeks of pregnancy
  pepsinogen-1 serum level was determined with blood samples taken from pregnant women with hyperemesis gravidarum and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Sevki Celen, MD, Study Chair — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data are available on request only due to ethical, legal or commercial reasons
Supporting Information: Analytic Code
Time Frame: two or three months

REFERENCES:
- [Result] Song M, Camargo MC, Weinstein SJ, Murphy G, Freedman ND, Koshiol J, Stolzenberg-Solomon RZ, Abnet CC, Mannisto S, Albanes D, Rabkin CS. Serum pepsinogen 1 and anti-Helicobacter pylori IgG antibodies as predictors of gastric cancer risk in Finnish males. Aliment Pharmacol Ther. 2018 Feb;47(4):494-503. doi: 10.1111/apt.14471. Epub 2017 Dec 15. PMID 29243850
- [Result] Han ML, Liou JM, Ser KH, Chen JC, Chen SC, Lee WJ. Changes of serum pepsinogen level and ABC classification after bariatric surgery. J Formos Med Assoc. 2021 Jun;120(6):1377-1385. doi: 10.1016/j.jfma.2020.10.029. Epub 2020 Nov 14. PMID 33199102
- [Result] Wei W, Zhang W, Li C, Kong H, Guo Z, Zhang Z, Bastien F, Gong Y, Wang H, Zhou L. Label-free detection of pepsinogen 1 and 2 by polyethylene coating Lamb microfluidic device. Biosens Bioelectron. 2019 Mar 15;129:231-237. doi: 10.1016/j.bios.2018.09.075. Epub 2018 Sep 21. PMID 30287174